CLINICAL TRIAL: NCT01009632
Title: Role of Exercise for Wound Healing in the Larynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Katherine Verdolini Abbott, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DC005643
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Acute Phonotrauma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Voice rest (Experimental)
  Interventions: Behavioral: Voice rest
- Resonant voice exercise (Experimental)
  Interventions: Behavioral: Resonant voice
- Spontaneous speech (Experimental)
  Interventions: Behavioral: Spontaneous speech

INTERVENTIONS:
Behavioral: Resonant voice — 4-hr of resonant voice exercise
  Arms: Resonant voice exercise
Behavioral: Voice rest — 4-hr of complete refrain from any voice use
  Arms: Voice rest
Behavioral: Spontaneous speech
  Other Names: 4-hr of conversational (normal) voice use
  Arms: Spontaneous speech

SUMMARY:
The purpose of this study is to explore quantitatively the hypothesis that "resonant voice," may enhance recovery from acute laryngeal phonotrauma, based on molecular assays from human laryngeal secretions and secondarily, clinical tests.

DETAILED DESCRIPTION:
The objective is to use the following operationalized question: Does a voicing mode shown to correspond to high-amplitude, low impact vocal cord oscillations, "resonant voice," improve the amount and time-course of recovery from acute phonotrauma, compared to vocal rest or spontaneous speech, as measured with molecular assays (primarily) and with behavioral and clinical tests (secondarily)?

ELIGIBILITY:
Inclusion Criteria:

* males and females who have had voice training and feel they are able to produce loud voice safely;
* ages 18-49;
* generally healthy;
* normal hearing bilaterally at 20 dB to 8,000 Hz; and
* demonstrated ability to produce "resonant voice" during training as determined by the examiner perceptually.

Exclusion Criteria:

* current chronic voice problems;
* current medications that are determined to possibly influence voice (e.g. diuretics, decongestants);
* heightened gag reflex;
* small nasal passage;
* deviated septum; and
* known or suspected allergy to anesthetics.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2004-02; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Biomarkers in laryngeal secretions | Up to 24-hour post-baseline

SECONDARY OUTCOMES:
Phonation Threshold Pressure (PTP) | Up to 24-hour post baseline
Direct Magnitude Estimations of phonatory effort (DME) | Up to 24-hour post baseline
Visual-perceptual ratings of the larynx | Up to 24-hour post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Verdolini Abbott, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Univesity of Pittsburgh, Pittsburgh, Pennsylvania, United States